CLINICAL TRIAL: NCT04387578
Title: Evaluation of Efficiency for Three Different Aligning Archwires During Initial Orthodontic Leveling: A Prospective Clinical Study
Brief Title: Evaluation of Efficiency for Three Different Aligning Archwires During Initial Orthodontic Leveling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Talaat Hussein Ali (Other)
Responsible Party: Sponsor-Investigator, Ahmed Talaat Hussein Ali, Principal Investigator, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 103
Record Dates: First submitted 2020-05-05; First posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Dental Malocclusion; Dental Crowding
Keywords: Orthodontic arch wire; alignment; Gummetal arch wire; multistrand arch wire
MeSH Terms: conditions — Malocclusion; Crowding | interventions — Orthodontic Appliances, Fixed

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A singlestrand NiTi arch wires (Experimental): in which 10 patients (5 males and 5 females) were treated with round singlestrand NiTi arch wires in a sequence of 0.012, 0.014, and 0.016 inch.
  Interventions: Device: fixed orthodontic appliance and arch wires
- Group B Gummetal arch wires (Experimental): in which 10patients (6 males and 4 females) were treated with niobium-titanium-tantalum-Zirconium arch wires (Gummetal arch wires) in a sequence of 0.014, 0.016, and 0.018 inch.
  Interventions: Device: fixed orthodontic appliance and arch wires
- Group C multistrand NiTi arch wires (Experimental): in which 10 patients (4males and 6females) were treated with multistrand NiTi arch wires in a sequence of 0.016, 0.018, and 0.020 inch.
  Interventions: Device: fixed orthodontic appliance and arch wires

INTERVENTIONS:
Device: fixed orthodontic appliance and arch wires — leveling and aligning stages in orthodontics

SUMMARY:
The present prospective clinical study was directed to evaluate the efficiency of three different aligning archwires during initial orthodontic leveling.

DETAILED DESCRIPTION:
The present prospective clinical study was directed to evaluate efficiency of three different aligning arch wires during initial orthodontic leveling.

The sample of present study included 30 patients, 15 females and 15 males; with a mean age was 17.81 ± 1.96 years. They were randomly allocated into three equal groups, according to the type of the aligning arch wire as follows:

1. Group A: in which 10 patients, with a mean age was 17.27 ± 1.95 years, were treated with conventional singlestrand NiTi arch wires.
2. Group B: in which 10 patients, with a mean age was 17.33 ± 2.42 years, were treated with Niobium-titanium-tantalum-Zirconium (Gummetal) arch wires.
3. Group C: in which 10 patients, with a mean age was 18.70 ± 1.49 years, were treated with multistrand NiTi arch wires.

Mandibular orthodontic study models were taken every 4 weeks and laser scanned to obtain 3D digital models during the 3 months observation period of the study. The changes in LII were determined at every 4 weeks observation intervals. Moreover, the changes in inter-canine, inter-1st premolar and inter-molar widths before and after three months were evaluated and compared among the three groups of aligning arch wires.

Data were collected and statistically analyzed via Statistical Package for Social Science (SPSS, version 23). One Way ANOVA and Kruskall-Wallis tests were used to assess the difference among the three studied groups and paired t-test was used to assess the difference and percent of changes within each group before and after three months observation period.

ELIGIBILITY:
Inclusion criteria:

* An age range from 15 to 20 years
* All permanent teeth have erupted (3rd molar not included)
* Angle class I malocclusion with normal facial proportions.
* Moderate crowding in the lower dental arch that required treatment with fixed appliance using the non-extraction approach.
* Good oral hygiene with healthy periodontium, good general health without any systematic disease that could affect the treatment.

Exclusion Criteria:

* Severe crowding that requires an extraction approach.
* A blocked-out tooth that prevent the easy placement of the bracket at the initial bonding appointment.
* Poor oral hygiene or periodontal compromised teeth.
* Relevant medical history and/or regular medication that contraindicates and/or interferes with orthodontic treatment.
* Craniofacial anomalies or previous history of trauma, bruxism, or parafunction.
* Previous orthodontic treatment.

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
evaluation of the alignment efficiency | three months of leveling and alignment
  evaluation of the alignment efficiency among the three investigated arch wires via the measurement of the scores of Little's Irregularity Index
comparison of the alignment efficiency | three months of leveling and alignment
  comparison of the alignment efficiency among the three investigated arch wiresvia the measurement of the scores of Little's Irregularity Index
evaluation of the alignment rate | three months of leveling and alignment
  evaluation of the alignment rate among the three investigated arch wiresvia the measurement of the scores of Little's Irregularity Index
comparison of the alignment rate among the three investigated arch wiresvia the measurement of the scores of Little's Irregularity Index | three months of leveling and alignment
  comparison of the alignment rate among the three investigated arch wiresvia the measurement of the scores of Little's Irregularity Index

SECONDARY OUTCOMES:
evaluation of the transverse mandibular arch dimensions changes among the three investigated arch wires. | three months of leveling and alignment
  evaluation of the transverse mandibular arch dimensions changes among the three investigated arch wires.
comparison of the transverse mandibular arch dimensions changes among the three investigated arch wires. | three months of leveling and alignment
  comparison of the transverse mandibular arch dimensions changes among the three investigated arch wires.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed T Ali, Demonstrator, Principal Investigator — Al-Azhar University
Locations (1):
- Al Azhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No